CLINICAL TRIAL: NCT03216044
Title: Incidence and Predictors of Chronic Pain After Vaginal Childbirth and C-section - a Prospective Cohort Study
Brief Title: Chronic Pain After Childbirth - Caesarean Section Compared to Vaginal Delivery and the Impact of Pre-existing Pain
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 451/2011BO2
Record Dates: First submitted 2017-06-28; First posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-01

CONDITIONS: Chronic Pain
Keywords: childbirth; caesarean delivery; vaginal delivery; chronic pain; painful sexual intercourse
MeSH Terms: conditions — Chronic Pain; Dyspareunia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is no doubt, that surgery is very often the beginning of a chronic pain disorder. C-section is a worldwide performed operation with increasing trend in the developed countries .This prospective cohort study evaluated the incidence of persistent pain after childbirth in respect of the pain status before childbirth and the modus of delivery.

DETAILED DESCRIPTION:
There are different variables that may influence the occurrence of chronic pain after childbirth. One of these could be c- section , pain status before childbirth or other psychological factors like fear of birth, irrational cognitive beliefs about delivery and perinatal complications. The pain status (intensity and location), demographic data, anesthesiological details and data about the circumstances of birth are evaluated by structured interview during pregnancy and 3 month and 12 moth after childbirth. The pregnant women received an individual code for access to the survey on the website of the study. The recruitment takes placed in doctors or midwifes office and by advertising. The commuting area was the city of Tuebingen (Germany). Women who feel uncomfortable with the media based survey supplied a written form. Study population is planned with 500 participants. The Institute for Clinical Epidemiology and Applied Biometry support the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* age of consent
* must be german-speaking

Exclusion Criteria:

- no written consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pregnant women living in the city of Tuebingen and Stuttgart or the area surrounding
Sampling Method: Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Incidence of new chronic pain disorder after vaginal delivery and after c-section | 3 months after delivery
  Surgery is often mentioned as cause of persistent postsurgical pain. C-section procedure could be related to the development of chronic pain after childbirth.
Incidence of new chronic pain disorder after vaginal delivery and after c-section | 12 month after delivery
  Surgery is often mentioned as cause of persistent postsurgical pain. C-section procedure could be related to the development of chronic pain after childbirth.

SECONDARY OUTCOMES:
Quality of Life (SF 12) after 12 months of delivery | 12 months after delivery
  The 12-Item Short Form Health Survey (SF-12) was developed for Medical Outcomes Study of patients with chronic conditions. Analysis of SF 12 in woman with chronic pain and without chronic pain after delivery

IPD SHARING:
Plan to Share IPD: No